CLINICAL TRIAL: NCT06958874
Title: Adjunctive Effect of Erythritol on Pocket Closure Rates: RCT
Brief Title: Adjunctive Effect of Erythritol on Pocket Closure Rates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, DDS, PhD, Associate Professor of Dentistry (PI), University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Verb n. 25 del 14/09/22 ABRUZZ
Record Dates: First submitted 2025-04-19; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Pocket, Periodontal; Pocket, Gingival
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Gingival Pocket

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSPT (Control) (Active Comparator): Participants receive standard non-surgical periodontal treatment (scaling and root planing) using ultrasonic and manual instruments in selected periodontal pockets.
  Interventions: Procedure: Non-surgical periodontal therapy alone
- NSPT + ERY (Test) (Experimental): Participants receive standard non-surgical periodontal treatment combined with sub-gingival air polishing using erythritol powder in selected periodontal pockets.
  Interventions: Procedure: Non-surgical periodontal therapy + sub-gingival air polishing

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy + sub-gingival air polishing — Participants receive a single session of non-surgical periodontal therapy (NSPT) using ultrasonic and manual instruments, combined with sub-gingival air polishing using erythritol powder. The treatment is applied to periodontal pockets with probing depth ≥ 4 mm in non-adjacent teeth.
  Arms: NSPT + ERY (Test)
Procedure: Non-surgical periodontal therapy alone — Participants receive a single session of non-surgical periodontal therapy (NSPT) using ultrasonic and manual instruments.
  Arms: NSPT (Control)

SUMMARY:
This clinical trial is studying whether using erythritol powder during non-surgical periodontal treatment (deep cleaning) helps improve gum health in people with severe periodontitis. Participants with deep gum pockets (4 mm or more) receive standard treatment alone or standard treatment plus cleaning with erythritol powder. The goal is to evaluate if adding erythritol improves outcomes such as healing of gum pockets, bleeding, plaque levels, and gum attachment compared to standard treatment alone.

DETAILED DESCRIPTION:
This study is testing whether erythritol powder, used during non-surgical periodontal treatment (also known as deep cleaning), can help improve gum health in people with advanced periodontitis (stage 3 or 4). Periodontitis is a serious gum infection that damages the soft tissue and bone supporting the teeth. Standard treatment includes removing plaque and tartar using manual tools or ultrasonic devices.

In this study, gum pockets that are 4 mm deep or more are treated either with standard care alone or with standard care plus a cleaning method that uses air pressure and erythritol powder (a sugar alcohol with antibacterial properties). The goal is to determine whether this additional step leads to improved clinical outcomes.

Participants are randomly assigned to one of the two treatments. The study tracks improvements in gum pocket depth after 2 and 4 months, as well as other indicators of periodontal health like bleeding and plaque levels. Researchers are also evaluating whether factors such as age, sex, smoking status, or diabetes influence treatment response.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older

Diagnosed with stage 3 or 4 periodontitis according to the 2017 classification

Presence of at least 12 natural teeth

Presence of periodontal pockets with probing depth ≥ 4 mm in non-adjacent teeth

Good general health or stable systemic conditions (e.g., controlled diabetes)

Exclusion Criteria:

Use of antibiotics or anti-inflammatory drugs within 3 months prior to treatment

Periodontal treatment in the previous 6 months

Pregnancy or breastfeeding

Current smokers of more than 10 cigarettes per day

Allergies or intolerance to erythritol or any materials used in the treatment

Systemic diseases or conditions that could influence periodontal healing (e.g., uncontrolled diabetes, immunodeficiency)

Use of medications known to affect periodontal tissues (e.g., phenytoin, cyclosporine, calcium channel blockers)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of periodontal pockets with successful pocket closure | 2 months and 4 months after treatment
  Percentage of treated periodontal pockets (with baseline probing depth ≥ 4 mm) that reach pocket closure, defined as probing pocket depth ≤ 4 mm without bleeding on probing, or ≤ 3 mm, at follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been determined whether individual participant data (IPD) will be shared. The decision will depend on institutional policies, data privacy considerations, and future research collaborations.